CLINICAL TRIAL: NCT05826093
Title: Cutaneous Sensory Block Area of the Subcostal Ultrasound-Guided Transversus Abdominis Plane Block
Acronym: CUSBAT
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSBA-SUSTAP
Record Dates: First submitted 2023-04-03; First posted 2023-04-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain
Keywords: Transversus abdominis plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients planned for cholecystectomy: Patients planned for elective laparoscopic cholecystectomy received a peroperative ultrasound-guided transversus abdominis plane (TAP) block at the beginning of the procedure.
  Interventions: Procedure: Ultrasound-guided subcostal transversus abdominis plane block (US-TAP)

INTERVENTIONS:
Procedure: Ultrasound-guided subcostal transversus abdominis plane block (US-TAP) — US-TAP is a peripheral nerve block applied for postoperative pain relief. Subcostal refers to the approach which can also be lateral or posterior. In this trial the subcostal approach was used.

SUMMARY:
Patients planned for elective laparoscopic cholecystectomy received a peroperative ultrasound-guided subcostal transversus abdominis plane block (USTAP) at the beginning of the procedure. At T90 minutes after the end of anaesthesia the cutaneous sensory block area (CSBA) was measured using cold sensation and mapped with a sterile marker. The CSBA was photodocumented and the area calculated.

ELIGIBILITY:
Inclusion Criteria:

* Planned for elective laparoscopic cholecystectomy, age 18 or older, written and verbal consent

Exclusion Criteria:

* Non-compliant due to language or psychiatric disease, previous surgery to the upper abdomen, incisional hernia, pregnancy, sensory deficit of the abdomen or thorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for elective laparoscopic cholecystectomy in a day surgery setting.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Cutaneous Sensory Block Area | 90 minutes postoperatively or 150 minutes after US-TAP application
  The area of the dermis which is blocked to sensory stimulus such as pain, heat and cold.

CONTACTS AND LOCATIONS:
Overall Officials: Cluas A Bertelsen, MD PhD, Study Chair — Copenhagen University Hospital - North Zealand
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salmonsen CB, Lange KHW, Rothe C, Kleif J, Bertelsen CA. Cutaneous sensory block area of the ultrasound-guided subcostal transversus abdominis plane block: an observational study. Reg Anesth Pain Med. 2024 Apr 2;49(4):289-292. doi: 10.1136/rapm-2023-104753. PMID 37640451